CLINICAL TRIAL: NCT01678196
Title: Helping Families Help Veterans With PTSD and Alcohol Abuse: An RCT of VA-CRAFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CRE 12-024
Record Dates: First submitted 2012-08-29; First posted 2012-09-03 (Estimated); Results first posted 2016-02-24 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-09

CONDITIONS: PTSD; Alcohol Abuse
Keywords: Family Members; Community Outreach; Internet
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- VA-CRAFT (Experimental): Family participants complete an on-line training course (VA-CRAFT) over a 3 month period
  Interventions: Behavioral: VA-CRAFT
- Control (Placebo Comparator): Participants will have the opportunity to complete the VA-CRAFT training program after 3 months; otherwise no intervention
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: VA-CRAFT — VA-CRAFT is an on-line training program that teaches family members how to communicate and interact with Veterans to promote their engagement in needed mental health services for PTSD or Alcohol Use Disorders. 12 on-line sessions.
  Arms: VA-CRAFT
Other: Control — Participants will have the opportunity to complete the VA-CRAFT training program after 3 months; otherwise no intervention
  Arms: Control

SUMMARY:
This project begins to evaluate the effectiveness of a web-based family outreach tool that is designed to promote treatment engagement among Veterans with posttraumatic stress disorder (PTSD) or alcohol use disorders (AUDs) but who have not yet engaged in mental health care. The National Center for PTSD has developed an on-line, Veteran-tailored, interactive web tool called VA - Community Reinforcement and Family Training (VA-CRAFT) that trains family members to effectively help their Veterans to engage in treatment for PTSD and/or AUDs. This project will provide preliminary information about VA-CRAFT's effectiveness.

DETAILED DESCRIPTION:
Background PTSD and AUDs are highly prevalent psychiatric disorders among combat Veterans that can lead to substantial impairments and disability. Although empirically supported treatments are available, the majority of Veterans suffering PTSD or AUDs do not engage in any mental health care. Data show that encouragement and support by family members play a key role in Veterans' willingness to engage in mental health care. However, many family members may not know how best to help their Veterans engage in mental health care. VA-CRAFT is an innovative adaptation of an empirically supported family training intervention (CRAFT) that has been shown to dramatically increase treatment engagement among substance abusing civilian samples. VA-CRAFT includes Veteran-specific content, a focus on PTSD, SUDs, or both, and also make use of interactive web-technology to increase its efficiency and reach. Pilot research is needed to begin to evaluate the effectiveness of this adaptation of an existing, efficacious intervention, to provide feedback to VA-CRAFT developers for possible modifications to content and delivery, and to inform future studies.

Objectives Specific aims are to: 1) provide pilot data on the effectiveness of VA-CRAFT on Veterans' mental health service utilization; 2) provide pilot data on the effectiveness of VA-CRAFT on family members' wellbeing, personal quality of life, perceived relationship quality with Veteran, and communication about treatment seeking; 3) obtain pilot data to explore possible differences in intervention response between Veterans with AUDs only, PTSD only, or both; and 4) provide information regarding potential changes in content and delivery as well as mediators and moderators of outcome for VA-CRAFT.

Methods This is a randomized controlled trial of VA-CRAFT that will obtain preliminary information on its effectiveness and pilot information to inform future studies. Participants will be drawn from a cohort of Veterans and family members enrolled in the Readiness and Resilience in National Guard Soldiers studies (RINGS; Polusny & Erbes, PIs). Using Veterans' responses to post-deployment RINGS surveys and administrative data, family members of Veterans who screen positive for PTSD or AUDs will be recruited and divided into 1 of 3 subsamples: 1) family of Veterans with AUDs only (anticipated n = 38), 2) family of Veterans with PTSD only (anticipated n = 72), and 3) family of Veterans with both PTSD and AUDs (anticipated n = 74; total anticipated N =184 across the 3 subsamples). Family member participants will complete baseline questionnaires of perceived Veteran PTSD and AUD symptoms, family functioning and communication, and well-being and will be randomly assigned to VA-CRAFT or Control (no treatment) conditions. Those assigned to the VA-CRAFT condition will complete the online VA-CRAFT course. Progress through VA-CRAFT will be monitored and stepped outreach efforts (emails, phone contacts) will be systematically used, as necessary, to promote completion of the intervention. Three months after the baseline assessment, family members and Veterans will complete follow-up questionnaires. Primary outcomes will include: 1) Veteran's mental health service utilization during the 3 months following initiation of VA-CRAFT as assessed by VA administrative data and 2) family member self-reports of wellbeing and quality of life and 3) family and Veteran reports of perceived relationship quality and communication about treatment seeking. Effect sizes will be estimated for each outcome within each subsample of participants (AUD only, PTSD only, and comorbid) and, if patterns are similar within subsamples, for the sample overall. Following the post-intervention questionnaires, qualitative interviews will be conducted with up to 40 family participants to examine possible moderators and mediators of treatment responses and to elicit participant feedback on VA-CRAFT modules and development to inform future VA-CRAFT development.

ELIGIBILITY:
Inclusion Criteria:

* Family participants:

  * must have participated in a Readiness and Resilience in National Guards Soldiers - (RINGS) study and be a spouse, partner, or family member of a Veteran who has also participated in a RINGS study
  * report frequent contact with the Veteran
  * be paired with a Veteran who has not received mental health services at VA or in the community for the past 3 months and who has screened positive for PTSD or AUDs
  * and have regular access to the internet.
* Veteran participants:

  * must have participated in a RINGS study
  * be in significant contact with a spouse/partner/family member who has enrolled in this protocol
  * screened positive for PTSD and/or AUD through their responses to a RINGS survey
  * and have not received mental health care (based on VA administrative data) or in the community for the past 3 months

Exclusion Criteria:

* Family members (and thus Veterans) will not be eligible for the study if they or their Veteran have reported severe levels of interpersonal violence in their relationship in the past 3 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2013-05; Primary Completion 2014-12 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher R. Erbes, PhD, Principal Investigator — Minneapolis VA Health Care System, Minneapolis, MN
Locations (1):
- Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tran T, Kuhn ER, Walser R, Drescher K. The relationship between religiosity, PTSD, and depressive symptoms in veterans in PTSD residential treatment. Journal of psychology and theology. 2012 Oct 1; 40(Winter 2012):313-322.
- [Background] Kuhn ER, Landes S. Mental and Behavioral Health Apps for Service Members, Veterans, and Providers. Society for Media Psychology & Technology: The Amplifier. 2013 Apr 1; Spring/Summer(2013):8-10.
- [Result] Reger GM, Hoffman J, Riggs D, Rothbaum BO, Ruzek J, Holloway KM, Kuhn E. The "PE coach" smartphone application: an innovative approach to improving implementation, fidelity, and homework adherence during prolonged exposure. Psychol Serv. 2013 Aug;10(3):342-349. doi: 10.1037/a0032774. PMID 23937084
- [Result] Erbes CR, Stinson R, Kuhn E, Polusny M, Urban J, Hoffman J, Ruzek JI, Stepnowsky C, Thorp SR. Access, utilization, and interest in mHealth applications among veterans receiving outpatient care for PTSD. Mil Med. 2014 Nov;179(11):1218-22. doi: 10.7205/MILMED-D-14-00014. PMID 25373044
- [Result] Kuhn E, Greene C, Hoffman J, Nguyen T, Wald L, Schmidt J, Ramsey KM, Ruzek J. Preliminary evaluation of PTSD Coach, a smartphone app for post-traumatic stress symptoms. Mil Med. 2014 Jan;179(1):12-8. doi: 10.7205/MILMED-D-13-00271. PMID 24402979
- [Result] Kuhn E, Eftekhari A, Hoffman JE, Crowley JJ, Ramsey KM, Reger GM, Ruzek JI. Clinician perceptions of using a smartphone app with prolonged exposure therapy. Adm Policy Ment Health. 2014 Nov;41(6):800-7. doi: 10.1007/s10488-013-0532-2. PMID 24398700
- [Result] Ruzek JI, Eftekhari A, Rosen CS, Crowley JJ, Kuhn E, Foa EB, Hembree EA, Karlin BE. Factors related to clinician attitudes toward prolonged exposure therapy for PTSD. J Trauma Stress. 2014 Aug;27(4):423-9. doi: 10.1002/jts.21945. PMID 25158635
- [Result] Whealin JM, Kuhn E, Pietrzak RH. Applying behavior change theory to technology promoting veteran mental health care seeking. Psychol Serv. 2014 Nov;11(4):486-94. doi: 10.1037/a0037232. PMID 25384001
- [Result] Owen JE, Jaworski BK, Kuhn E, Makin-Byrd KN, Ramsey KM, Hoffman JE. mHealth in the Wild: Using Novel Data to Examine the Reach, Use, and Impact of PTSD Coach. JMIR Ment Health. 2015 Mar 25;2(1):e7. doi: 10.2196/mental.3935. eCollection 2015 Jan-Mar. PMID 26543913
- [Result] Williams EC, Gupta S, Rubinsky AD, Jones-Webb R, Bensley KM, Young JP, Hagedorn H, Gifford E, Harris AH. Racial/Ethnic Differences in the Prevalence of Clinically Recognized Alcohol Use Disorders Among Patients from the U.S. Veterans Health Administration. Alcohol Clin Exp Res. 2016 Feb;40(2):359-66. doi: 10.1111/acer.12950. PMID 26842254

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were partners of Veterans who had screened positive for PTSD or alcohol use disorders in prior surveys with the study team. Of 287 identified eligible partners, 190 were successfully reached and 66 consented to be in the study.
Period: Overall Study
Arm/Group | VA-CRAFT | Control
Started | 34 | 32
Completed | 34 (Primary outcome data was from the electronic medical record and was available for all participants.) | 32 (Primary outcome data was from the electronic medical record and was available for all participants.)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VA-CRAFT | Control | Total
Number analyzed (Participants) | 34 | 32 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 32 | 66
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 32 | 66
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 21 | 21 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 13 | 10 | 23
Region of Enrollment [Number; unit: participants]
  United States | 34 | 32 | 66

OUTCOME MEASURES:

1. Primary Outcome: Veteran Engagement in VA Mental Health Services
Description: Administrative data on mental health service utilization for Veterans will be compared for those whose family members receive the intervention (VA-CRAFT) and those who do not.
Time Frame: 3 months after initiation of the intervention
Measure: Number; unit: participants
Arm/Group | VA-CRAFT | Control
Number analyzed (Participants) | 34 | 32
participants | 4 | 4
Statistical Analysis 1: Comparison: VA-CRAFT vs Control; Test type: Superiority or Other; p = 0.927, Chi-squared

2. Secondary Outcome: Family Member Psychosocial Wellbeing: Brief Symptom Inventory - 18
Description: Brief Symptom Inventory - 18 (Derogatis, 1993) is an 18 item measure of general mental health symptoms and distress. The total score is used, which is the mean of 18 items rated from 0 (not at all) to 4 (extremely) distressing. Total scores range from 0 (low distress) to 4 (high distress).
Time Frame: 3 months after initiation of the intervention
Population: Group sample sizes are smaller than total sample sizes due to missing data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | VA-CRAFT | Control
Number analyzed (Participants) | 32 | 29
units on a scale | 0.46 (0.52) | 0.58 (0.59)
Statistical Analysis 1: Comparison: VA-CRAFT vs Control; Test type: Superiority or Other; p = 0.67, ANCOVA; ANCOVA reflects change from Time 1 scores (entered as covariate) to Time 2 Scores

3. Secondary Outcome: Family Functioning
Description: Relationship Happiness Scale. The RHS is a 9 item scale of general happiness in close relationships. The total score is reported here, reflecting the mean of the 9 items rated on a scale of 1 (completely unhappy) to 10 (completely happy). Higher total scores reflect greater relationship happiness.
Time Frame: 3 months after the initiation of the intervention
Population: Sample sizes are smaller than the overall sample due to missing questionnaire data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | VA-CRAFT | Control
Number analyzed (Participants) | 32 | 28
units on a scale | 5.92 (1.78) | 5.75 (2.36)
Statistical Analysis 1: Comparison: VA-CRAFT vs Control; Test type: Superiority or Other; p = 0.743, ANCOVA; ANCOVA results include Time 1 scores as a covariate, thus reflecting change over time

4. Secondary Outcome: Caregiver Burden
Description: Caregiver Burden Scale (CBS). The CBS is a 16 items scale assessing caregiver burden. It has 16 items rated from 1 (not at all) to 5 (extremely) distressed or burdened. Scores reported are the total scale scores, calculated as the mean of the 16 items, with a range from 1 (low burden) to 5 (high burden).
Time Frame: 3 months post-randomization
Population: Sample sizes are smaller than total sample size due to missing questionnaire data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | VA-CRAFT | Control
Number analyzed (Participants) | 32 | 29
units on a scale | 1.56 (0.49) | 1.84 (0.88)
Statistical Analysis 1: Comparison: VA-CRAFT vs Control; Test type: Superiority or Other; p < .001, ANCOVA; ANCOVA reflects change for Time 1 values (entered as the covariate) to Time 2 values (entered as the DV)

ADVERSE EVENTS:
Arm/Group | VA-CRAFT | Control
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/32
Other Adverse Events (participants affected / at risk) | 0/34 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No